CLINICAL TRIAL: NCT01257906
Title: A MULTICENTER, DOUBLE-BLIND, RANDOMIZED, VEHICLE-CONTROLLED, PARALLEL-GROUP STUDY COMPARING CLINDAMYCIN PHOSPHATE (1.2%) AND TRETINOIN (0.025%) TOPICAL GEL (ACTAVIS MID-ATLANTIC LLC) TO ZIANA® (CLINDAMYCIN PHOSPHATE 1.2% AND TRETINOIN 0.025%) GEL (MEDICIS, THE DERMATOLOGY COMPANY®) AND BOTH ACTIVE TREATMENTS TO CLINDAMYCIN PHOSPHATE (1.2%) AND TRETINOIN (0.025%) TOPICAL GEL PLACEBO (ACTAVIS MID-ATLANTIC LLC) IN THE TREATMENT OF MILD TO SEVERE ACNE VULGARIS
Brief Title: Bioequivalence Study Comparing Clindamycin Phosphate (1.2%) and Tretinoin (0.025%) Topical Gel to Ziana and Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Actavis Mid-Atlantic LLC (Industry)
Responsible Party: Christine M. Winslow, Ph.D., Director Clinical Development, Actavis Mid-Atlantic LLC
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Acta/Clin-Tret/2009
Record Dates: First submitted 2010-12-09; First posted 2010-12-10 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2010-12

CONDITIONS: MILD TO SEVERE ACNE VULGARIS
Keywords: acne; Ziana; clindamycin; tretinoin
MeSH Terms: conditions — Acne Vulgaris | interventions — Tretinoin; Gels; clindamycin, tretinoin drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CLIND PHOSPHATE (1.2%) AND TRETINOIN (0.025%) TOPICAL GEL (Experimental): Topical Gel Test Product
  Interventions: Drug: CLIND PHOSPHATE (1.2%) AND TRETINOIN (0.025%) TOPICAL GEL
- ZIANA® (Active Comparator): Topical Gel Reference Product
  Interventions: Drug: ZIANA®
- Vehicle Control (Placebo Comparator): Topical Gel Placebo
  Interventions: Drug: Vehicle Control

INTERVENTIONS:
Drug: CLIND PHOSPHATE (1.2%) AND TRETINOIN (0.025%) TOPICAL GEL — Topical Gel applied in the evening for 84 days
  Arms: CLIND PHOSPHATE (1.2%) AND TRETINOIN (0.025%) TOPICAL GEL
Drug: ZIANA® — Topical Gel applied in the evening for 84 days
  Arms: ZIANA®
Drug: Vehicle Control — Topical Gel applied in the evening for 84 days.
  Arms: Vehicle Control

SUMMARY:
ZIANA® (clindamycin phosphate 1.2% and tretinoin 0.025%) gel, marketed by Medicis, The Dermatology Company®, is a safe and effective topical therapy used for the treatment of acne vulgaris. Actavis Mid-Atlantic LLC has developed a generic formulation of clindamycin phosphate (1.2%) and tretinoin (0.025%) topical gel and the current study is designed to evaluate the bioequivalence of this formulation to ZIANA®.

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant female patients must be between the ages of 12 and 40 years old inclusive. 2. Patients who are 18 years of age or older must have provided IRB/IEC approved written informed consent. Patients between the ages of 12 to 17 years of age must have provided IRB/IEC approved written assent; this written assent must be accompanied by an IRB/IEC approved written informed consent from the patient's legally acceptable representative (i.e., parent or guardian). In addition, all patients or their legally acceptable representatives (i.e., parent or guardian) must sign a HIPAA authorization, if applicable. 3. Patients must have a definite clinical diagnosis of mild to severe acne vulgaris (Grade 2, Grade 3 or Grade 4 on the IGE). 4. Patients must have a minimum of 20 and a maximum of 100 facial inflammatory lesions at baseline. Patients must also have a minimum of 25 and a maximum of 100 non-inflammatory lesions (i.e., open and closed comedones) at baseline. Patients may have no more than two (2) nodulo-cystic lesions at baseline. For the purposes of study treatment and evaluation, these lesions should be limited to the facial treatment area. Lesions involving the eyes, angles of the nose (i.e., the lines around your nostrils and under the nostrils) and scalp should be excluded from the count. Patients may have acne lesions on other areas of the body (e.g., on the back). 5.Female patients of childbearing potential must have been using accepted methods of birth control or must agree to continue to practice abstinence, from 30 days prior to study entry to 30 days after the last administration of study drug. All female patients are considered to be of childbearing potential unless they have been surgically sterilized or have been postmenopausal for at least 1 year. Abstinence is an acceptable method of birth control. Alternatively, any of the following methods of birth control are acceptable: oral contraceptives, contraceptive patches/implants (e.g., Norplant®) Depo-Provera®, double barrier methods (e.g., condom and spermicide) or IUD. Female patients must have a negative urine pregnancy test at baseline. A negative result of a pregnancy test having a minimum sensitivity of at least 50 mIU/ml for hCG should be obtained. 6. All male patients must agree to use accepted methods of birth control with their partners, from the day of the first dose administration to 30 days after the last administration of study drug. Abstinence is an acceptable method of birth control. Alternatively, any of the following methods of birth control are acceptable: oral contraceptives, contraceptive patches/implants (e.g., Norplant®), Depo-Provera®, double barrier methods (e.g., condom and spermicide) or IUD. 7. Patients must be willing and able to understand and comply with the requirements of the protocol, including attendance at the required study visits. 8. Patients must be willing to refrain from using any treatments for acne vulgaris, including antibiotics, other than the investigational product, for acne present on the face. Patients may use other topical acne treatments that do not have significant or measurable systemic absorption for treatment of acne of the back, shoulders and chest (e.g., benzoyl peroxide, salicylic acid). 9. Patients must be in good health and free from any clinically significant disease. 10. Patients who use make-up must have used the same brands/types of make-up for a minimum period of 14 days prior to study entry and must agree to not change make-up brand/type or frequency of use throughout the study.

Exclusion Criteria:

1. Female patients who are pregnant, nursing or planning to become pregnant during study participation (Visit 1 through Visit 5) will be excluded from study participation. 2. Patients who have a known hypersensitivity to clindamycin phosphate or tretinoin or their excipients will be excluded from study participation. 3. Patients who have conditions that may interfere with the evaluation of acne vulgaris. Such conditions include, but are not limited to the following: rosacea; seborrheic dermatitis; perioral dermatitis; corticosteroid-induced acne or folliculitis; carcinoid syndrome; squamous cell carcinoma; mastocytosis; acneiform eruptions caused by make-up or medication; bacterial folliculitis; facial psoriasis; and facial eczema. 4. Patients who have acne congoblata, acne fulminans, and secondary acne (e.g., chloracne and drug induced acne) will be excluded from participation. 5. Patients who have been treated with systemic antibiotics or systemic anti-acne drugs or systemic anti-inflammatory drugs within 30 days prior to baseline will be excluded from study participation. 6. Patients who have been treated with prescription and/or over-the-counter topical medications for the treatment of acne vulgaris including antibiotics, topical corticosteroids,,α-hydroxy/glycolic acid, benzoyl peroxide, or topical anti-inflammatory medications on the face within 14 days prior to baseline will be excluded from study participation. 7. Patients who have used erythromycin or erythromycin containing products in any form within 30 days prior to study entry (i.e., Visit 1) will be excluded from study participation. 8. Patients who are currently taking or have been treated with corticosteroids (including intranasal and inhaled corticosteroids) within 30 days prior to baseline will be excluded from study participation. 9. Patients who have started hormonal therapy or changed the dosage of their hormonal therapy within 3 months prior to baseline will be excluded from study participation. The dosage and frequency of use of any hormonal therapy started greater than 3 months prior to baseline must remain unchanged throughout the study (Visit 1 through Visit 5). Hormonal treatments include, but are not limited to, estrogenic and progestational agents such as birth control pills. 10. Patients who use androgen receptor blockers for acne (such as spironolactone or flutamide) will be excluded from study participation. 11. Patients who have received oral retinoids (e.g., isotretinoin) within 180 days prior to study entry,or have used therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed) within 180 days prior to study entry, or have applied topical retinoids (e.g., tretinoin, tazarotene, adapalene) to the face within the 30 days prior to baseline will be excluded from study participation. 12. Patients who have received radiation therapy and/or anti-neoplastic agents within 90 days prior to baseline will be excluded from study participation. 13. Patients who have unstable medical disorders that are clinically significant or life-threatening diseases will be excluded from study participation. 14. Patients who have on-going malignancies requiring systemic treatment will be excluded from study participation. In addition, patients who have any malignancy of the skin of the facial area will be excluded from study participation. 15. Patients who have facial hair will be excluded from study participation. Unacceptable facial hair includes, but is not limited to, beards, and long side-burns. A well-trimmed mustache is acceptable. Patients who have performed wax epilation of the face within 14 days prior to baseline will also be excluded from study participation. 16. Patients who engage in activities that involve excessive or prolonged exposure to sunlight or weather extremes, such as wind or cold, will be excluded from study participation. 17. Patients who consume excessive amounts of alcohol (greater than two drinks per day) or use drugs of abuse (including, but not limited to, cannabinoids and cocaine) as judged by history will be excluded from study participation. 18. Patients who have participated in an investigational drug study (i.e., patients have been treated with an investigational drug) within 30 days prior to baseline will be excluded from study participation. Patients who are participating in non-treatment studies such as observational studies or registry studies can be considered for inclusion. 19. Patients who have been previously enrolled in this study will be excluded from study participation. 20. Patients who have had within 30 days prior to baseline or during the study cryodestruction or chemodestruction, dermabrasion, photodynamic therapy, acne surgery, intralesional steroids, or x-ray therapy will be excluded from study participation. 21. Patients who have had laser therapy, and electrodesiccation to the facial area within 180 days prior to study entry will be excluded from participation. 22. Patients who have had cosmetic procedures (e.g., facials) which may affect the efficacy and safety profile of the investigational product within 14 days prior to study entry will be excluded from participation. 23. Patients who have had general anesthesia for any reason and patients who have received neuromuscular blocking agents within 14 days prior to study entry will be excluded from study participation. 24. Patients who have a history of Crohn's disease, ulcerative colitis, regional enteritis, antibiotic-associated colitis will be excluded from study participation. 25. Patients who have a baseline local irritation score of 3 (severe, marked/intense) as scored using the Application Site Reaction Scale (Section 5.2) will be excluded from participation.

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1225 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Therapeutic Equivalence | 12-weeks
  The primary equivalence comparison is that between the test and reference products for the mean percent change from baseline in the inflammatory lesion counts and the non-inflammatory lesion counts at Visit 5.
Superiority | 12-Weeks
  The primary superiority evaluations are the comparisons between each active treatment and the vehicle control relative to the mean percent change in the inflammatory lesion counts and the non-inflammatory lesion counts.
Safety | 12-Weeks
  All treatment-emergent adverse events reported during the study will be summarized in order to assess safety.

CONTACTS AND LOCATIONS:
Overall Officials: Madhuri Tadepalli, MD, Principal Investigator — Skin and Cosmetology Clinic; Bela J. Shah, MD, Principal Investigator — BJ Medical College and Civil Hospital; Abir Saraswat, MD, Principal Investigator — Indu Shree Clinic; Manoj K. Parekh, MD, Principal Investigator — Bhagwan Mahaveer Jain Hospital; V. R. Sardesai, MD, Principal Investigator — Sardesai Clinic; Girish BS, MD, Principal Investigator — Justice KS Hedge Charitable Hospital; Leelavathy B., MD, Principal Investigator — Bowring & Lady Curzon Hospital; Rajkumar V., MD, Principal Investigator — Dhanawantari Polyclinic; Mukta Sachdev, MD, Principal Investigator — MS Clinical Research Pvt. Ltd; Anilkumar Malik, MD, Principal Investigator — G.M Modi Hospital; Narayana Rao, MD, Principal Investigator — Skin and Cosmetology; Guru Prasad, MD, Principal Investigator — Dayal Clinic; Jayadev Betkerur, MD, Principal Investigator — J.S.S. Medical College Hospital; Bhanuja Rani, MD, Principal Investigator — GVK Clinic; Mishra RS, MD, Principal Investigator — Skin Care and Cosmetology Centre; Hemanji R. Jerajani, MD, Principal Investigator — L.T.M. Medical College & General Hospital; BV Ramachandra, MD, Principal Investigator — Andhra Medical College; Akhilesh Agarwal, MD, Principal Investigator — Twacha Skin and Hair Clinic; Deepak Kotkar, MD, Principal Investigator — Dr. Deepak Kotkar Clinic; Alur S. Kumar, MD, Principal Investigator — Owaisi Hospital & Research Centre; Jayesh Kothari, MD, Principal Investigator — Skin Clinic; MG Gopal, MD, Principal Investigator — Kempegowda Institute of Medical Sciences; D. N. Balraj, MD, Principal Investigator — Rajbal Skin Clinic; Meethesh Agrawal, MD, Principal Investigator — Skin Clinic; Ravi M. Rathod, MD, Principal Investigator — Skin Care Centre; Ranjan C. Raval, MD, Principal Investigator — Smt. NHL Medical College and V.S. Hospital; V. K. Somani, MD, Principal Investigator — Somani Skin and Cosmetology Institute; Kailash Bhatia, MD, Principal Investigator — Bhatia Skin, Laser, & Cosmetic Center; Bhavesh K. Swarnakar, MD, Principal Investigator — Swarnakar's Clinic; Jayakar Thomas, MD, Principal Investigator — J.T. Skin Care Centre; Karigi Siddalingappa, MD, Principal Investigator — Vijayanagara Institute Of Medical Sciences; DVS Pratap, MD, Principal Investigator — Durga Bai Deshmukh Hospital and Research Center; Amit Madan, MD, Principal Investigator — Madan's Skin Care Centre; Rajeev Agarwal, MD, Principal Investigator — MV Hospital and Research Center; Ramesh Bhat, MD, Principal Investigator — Father Muller Medical College and Hospital; Ravindra B P, MD, Principal Investigator — Raga's Skin Care; S. Sacchidananda, MD, Principal Investigator — CITI Hospital; Veena Patil, MD, Principal Investigator — Medi Derma Hospital; Dinesh V Deshpande, MD, Principal Investigator — Deshpande Skin Clinic; Ajay J Deshpande, MD, Principal Investigator — Dr. Ajay Deshpande's Clinic; Sudhakar Grandhi, MD, Principal Investigator — Medipoint Hospitals Pvt. Ltd.; Anirudh D. Gulanikar, MD, Principal Investigator — Gulanikar Skin Clinic; Prashant K Palwade, MD, Principal Investigator — Keshav Skin and Hair Clinic; Uday Kulkarni, MD, Principal Investigator — Skin Care and Cosmetology Clinic; Amit Luthra, MD, Principal Investigator — Ishira Skin Clinic; K Venkatachalam, MD, Principal Investigator — Sri Gayathri Skin Care and Hair Transplant Centre; Apoorva Jain, MD, Principal Investigator — Max Skin Care Centre; Pradyumna P Vaidya, MD, Principal Investigator — Clinical Development Centre Pvt. Ltd.; Prachi A Matte, MD, Principal Investigator — Derma Lazer Clinic; Vikrant A Saoji, MD, Principal Investigator — Dr. Vikrant Saoji Skin Clinic; Archana M Goyal, MD, Principal Investigator — Laser and Skin Clinic Jaipur; Anshu Jain, MD, Principal Investigator — Skin Clinic; Vijay Zawar, MD, Principal Investigator — Skin Clinic; Sushil Y Pande, MD, Principal Investigator — Sparsh Hospital and Poly Clinic; Sujata Sengupta, MD, Principal Investigator — BP Poddar Hospital and Medical Research Limited; Kote R Purushottam, MD, Principal Investigator — Skin Care Clinic; Kiran Godse, MD, Principal Investigator — Shree Skin Centre and Pathology Laboratory
Locations (1):
- Lotus Labs Pvt. Ltd, Bangalore, India